CLINICAL TRIAL: NCT01316770
Title: A Randomized Within-Subject, Double-Blind, Placebo-Controlled Study of Dexamethasone Irrigation of the Parotid Glands in Primary Sjögren's Syndrome Subjects
Brief Title: Dexamethasone Irrigation of the Parotid Glands in Primary Sjögren's Syndrome Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 110094; 11-D-0094 (Other: CNS IRB number)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Sjögren's Syndrome; Xerostomia
Keywords: Xerostomia; Sjögren's Syndrome; Interventional Study; Sjogren's Syndrome; Dry Mouth
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Parotid Irrigation (Placebo Comparator): Within-Subject, Double-Blind, Placebo-Controlled Study. This parotid gland is irrigated with saline (placebo). { UPDATE: drug(generic) was administered at what time pt, dose of drug, route administration, frequency}
  Interventions: Drug: Placebo Parotid Irrigation
- Dexamethasone Parotid Irrigation (Experimental): Within-Subject, Double-Blind, Placebo-Controlled Study. This parotid gland is irrigated with dexamethasone {UPDATE: drug (generic) was administered at what time pt, dose of drug, route administration, frequency}
  Interventions: Drug: Dexamethasone Parotid Irrigation

INTERVENTIONS:
Drug: Dexamethasone Parotid Irrigation — Irrigation of the parotid gland from one side of the mouth with dexamethasone.
  Other Names: Placebo Parotid Irrigation
  Arms: Dexamethasone Parotid Irrigation
Drug: Placebo Parotid Irrigation — Irrigation of the parotid gland on the opposite side of the mouth with placebo saline.
  Arms: Placebo Parotid Irrigation

SUMMARY:
Background:

Sjögren's syndrome is an autoimmune disease (where the immune system attacks normal body tissues) that affects the salivary glands. Many people with Sjögren's syndrome are not able to make enough saliva because their salivary glands are inflamed. The dry mouth that results can interfere with daily activities and can lead to dental cavities, mouth sores, and infections. Injections of corticosteroids into the parotid glands can improve saliva production in people with Sjögren's syndrome, but current treatment practices may provide only temporary relief. Researchers are interested in studying the effectiveness of stronger corticosteroid injections (using dexamethasone) to determine how the corticosteroid treatment actually works.

Objectives:

- To evaluate the effectiveness and mechanics of dexamethasone injections to improve saliva production in individuals with primary Sjögren's syndrome.

Eligibility:

- Women between 18 and greater of age who have been diagnosed with primary Sjögren's syndrome, and have had a biopsy of the minor salivary glands in the past 5 years that shows a moderate level of inflammation.

Design:

* Participants will be screened with a full medical history and physical examination, blood and urine tests, and salivary gland biopsies. Participants will also be screened with tests of saliva flow production and evaluation of the salivary ducts and glands, and will complete questionnaires about dry mouth symptoms.
* At the first treatment visit, participants will receive an injection of dexamethasone into one parotid gland and an injection of saline into the other gland. After the injections, participants will provide a blood sample to test the level of dexamethasone in the blood.
* Two weeks after the first treatment, participants will return for an evaluation visit to have saliva flow rate measurements taken, and will complete a questionnaire about dry mouth symptoms.
* Four weeks after the first treatment, participants will have a second treatment for each parotid gland, with the same tests and questionnaires as before.
* Participants will have additional evaluation visits 6 and 8 weeks after the first treatment visit, with a followup telephone call approximately 6 weeks after the last dexamethasone treatment visit.

DETAILED DESCRIPTION:
BACKGROUND:

Salivary gland dysfunction is one of the major manifestations of Sjögren's (SS). Although inflammation is thought to play an important role in the exocrinopathy, the correlation between glandular dysfunction and inflammation is limited. Systemic anti-inflammatory therapies tested to date, such as tumor necrosis factor antagonists, have not been effective treatments for SS salivary hypofunction, raising doubts about inflammation being the sole cause of salivary gland dysfunction. However, none of these trials tested whether an anti-inflammatory effect was achieved in glandular tissues.

Studies by Izumi et al found that a limited course of low-dose topical corticosteroid applied to the parotid glands resulted in sustained improvement in saliva production. Unfortunately, these studies did not examine the mechanistic effects of corticosteroids on the major salivary glands. A plausible assumption is that corticosteroids improved salivary gland function by reducing inflammation, although other or associated mechanisms, such as an improved transcellular ion transport in epithelial cells cannot be ruled out. This study aims to study the efficacy of low-dose topical corticosteroid (dexamethasone) irrigation of the parotid gland in reducing salivary dysfunction in subjects with SS, and also to evaluate the effects of treatment on inflammation and other possible mechanistic processes.

PRIMARY OBJECTIVE:

- To determine whether irrigation of the parotid gland with low-dose topical dexamethasone improves parotid salivary gland flow in SS subjects.

SECONDARY OBJECTIVES:

* To perform mechanistic studies to determine the mechanisms of action of low-dose topical corticosteroid irrigation of the parotid gland.
* To assess biomarkers of inflammation and salivary gland dysfunction in SS subjects treated with low-dose topical corticosteroid irrigation of the parotid glands.
* To assess localized safety of dexamethasone irrigation of the parotid gland, as compared with placebo.

STUDY POPULATION:

The study will enroll up to 20 adult females with primary SS in order to randomize and treat 16 subjects. Key enrollment criterion include a focus score of greater than or equal to 3 on minor salivary gland biopsy in the previous 5 years and measurable stimulated bilateral parotid salivary flow (greater than or equal to 0.01 mL/min per gland). Subjects will be recruited from protocol 84-D-0056, conducted at the National Institutes of Health (NIH).

DESIGN:

This will be a single-site, randomized-within-subject, double-blind, placebo-controlled, phase 2 pilot study in which all subjects receive both active drug (dexamethasone) and placebo (normal saline), thereby acting as their own controls.The study design is doubly-repeated measures; within a subject, measures are repeated in both time and treatment (i.e., one side of mouth receives dexamethasone while the other receives placebo.). After baseline assessment of salivary flow and other measurements of salivary function, subjects will be randomly assigned, in a double-blind fashion, to dexamethasone irrigation of one parotid gland and normal saline irrigation of the other parotid gland. They will undergo a total of 2 treatment sessions, 4 weeks apart (Days 0 and 28). Post-treatment assessments of salivary flow, dry mouth symptoms, and adverse events (AEs) will be performed at specified intervals.

OUTCOME MEASURES:

Primary Endpoint:

- Change in salivary flow from Day 0 to Day 56.

Secondary Endpoints:

* Change in focus score on parotid biopsy from Screening to Day 56.
* Change in salivary flow from Day 0 to study Days 14, 28, 42, and 56.
* Changes in assessments on the Patient Dry Mouth Questionnaire from Day 0 to study Days 14, 28, 42, and 56.
* Changes in assessments on the Sj(SqrRoot)(Delta)gren s Disease Activity Index from Day 0 to study Days 14, 28, 42, and 56.
* Changes in other assessments of salivary function from baseline to study Day 56, including technetium scan of the salivary glands.
* Changes in laboratory measures of inflammation.
* Frequency of AEs related to treatment; AE location (body site, right or left), will be recorded and evaluated, as applicable.

Exploratory endpoints

- Changes in mechanistic endpoints from baseline to study Days 14, 28, 42, and 56.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Female gender and age 18 and greater.
* Diagnosed with primary SS in Protocol 84-D-0056.
* Stimulated salivary flow of at least 0.01 mL/min from each parotid gland, using the standard operating procedure (SOP) for the National Institute of Dental and Craniofacial Research (NIDCR) Molecular Physiology and Therapeutics Branch (MPTB) Sjögren's Syndrome Clinic
* Minor salivary gland (MSG) biopsy with a focus score of greater than or equal to 1 obtained 0 to 7 years prior to study enrollment. Biopsies from outside of the National Institutes of Health (NIH) must be reviewed by the NIH Pathology Department. An MSG biopsy will be required for the following situations:
* The last biopsy was obtained before the use of rituximab.
* The last biopsy was obtained before the use of immunosuppressants, biologics, or disease-modifying antirheumatic drugs for more than 3 months.
* The last biopsy was obtained before the use of systemic corticosteroids (for more than 2 weeks or for shorter periods at doses of more than 0.5 mg/kg) or local parotid corticosteroids. The use of topical or intra-articular/periarticular corticosteroids will not require a repeat biopsy.
* For women of childbearing potential, use of, or willingness to use, an effective method of birth control during the study. Effective methods include abstinence, history of hysterectomy, tubal ligation, intrauterine device, licensed hormonal methods, condoms, diaphragm, and cervical cap.
* Ability to provide written informed consent prior to entry in the study.

EXCLUSION CRITERIA:

* History of lymphoma.
* History of mycosis, aspergillosis, or other deep fungal infection of the parotid gland.
* History of salivary gland malignancy (primary or metastatic to the salivary gland).
* History of secondary Sjögren's syndrome.
* Parotid infection that does not resolve at least 4 weeks before the start of the Screening Period.
* Any active viral infection that does not resolve by the start of the Screening Period.
* Pregnancy or lactation.
* Use of biologics within 3 months of the start of the Screening Period.
* Any experimental therapy within 3 months before the start of the Screening Period.
* Use of immunosuppressants such as methotrexate, leflunomide, azathioprine, cyclophosphamide, systemic cyclosporine, or systemic corticosteroids within 3 months prior to the start of the Screening Period.
* Use of inhaled corticosteroids within 3 months prior to the start of the Screening Period.
* Use of antimalarials and regular use of NSAIDs unless the dose has been stable (or decreased) for at least 2 months.
* Inability to discontinue the use of saliva stimulants such as pilocarpine and cevimeline for 24 hours before each study visit.
* Parotid intraductal irrigation or instillation with steroids within the past year.
* Use of rituximab within 6 months prior to the start of the Screening Period.
* Allergy to steroids or technetium, or any components of the formulations.
* Current use of warfarin or heparin.
* History of bleeding disorder.
* Both severe atrophy and fibrosis of the MSG noted on the pathology report of the MSG biopsy.
* Inability to comply with protocol procedures and the number of required visits.
* Inability to cannulate one or both parotid glands.
* Parotid fill volume less than 0.5 mL in one or both parotid glands.
* Significant concurrent medical condition or other circumstances that, in the opinion of the principal investigator, could affect the subject's ability to tolerate or complete the study.
* Unable to understand written English for completion of study questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05-01; Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilias G Alevizos, D.M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Izumi M, Eguchi K, Nakamura H, Takagi Y, Kawabe Y, Nakamura T. Corticosteroid irrigation of parotid gland for treatment of xerostomia in patients with Sjogren's syndrome. Ann Rheum Dis. 1998 Aug;57(8):464-9. doi: 10.1136/ard.57.8.464. PMID 9797551
- [Background] Takagi Y, Katayama I, Tashiro S, Nakamura T. Parotid irrigation and cevimeline gargle for treatment of xerostomia in Sjogren's syndrome. J Rheumatol. 2008 Nov;35(11):2289-91. doi: 10.3899/jrheum.080370. No abstract available. PMID 19004065
- [Background] Manor W. A clinical learning experience in discharge planning. Nurse Educ. 1991 Nov-Dec;16(6):35. No abstract available. PMID 1754137
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-D-0094.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants were screened in the United States. Nine of the participants were then eligible and enrolled between October, 2011 and Sep, 2013 and administered treatment.
Pre-assignment Details: Screening occurred in two stages: Stage I (within 6 weeks before Stage II), and Stage II (within 6 weeks before randomization). Ten participants were eligible following the Stage I screening, but one subject loss their eligibility at Stage II screening because she refused the parotid biopsy.
Units Other Than Participants: parotid glands
Groups:
- Dexamethasone Irrigation of Parotid Gland: Parotid salivary gland on the side of the mouth that received dexamethasone irrigation on study Day 0 and study Day 28.
- Placebo Irrigation of Parotid Gland: Parotid salivary gland on the side of the mouth that received placebo irrigation on study Day 0 and study Day 28.
Period: Overall Study
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Started | 9; 9 parotid glands (Each study participant received the dexamethasone parotid irrigation on one side of mouth.) | 9; 9 parotid glands (Each study participant received the placebo parotid irrigation on the other side of mouth.)
Completed | 9; 9 parotid glands | 9; 9 parotid glands
Not Completed | 0; 0 parotid glands | 0; 0 parotid glands

BASELINE CHARACTERISTICS:
Population: Safety Population: all enrolled participants that received any parotid saline irrigation used to determine parotid filling volume during Stage I screening.
Units Other Than Participants: parotid glands
Groups:
- Overall Study: Safety Population: all enrolled participants that received any parotid saline irrigation used to determine parotid filling volume during Stage I screening.
Arm/Group | Overall Study
Number analyzed (Participants) | 11
Number analyzed (parotid glands) | 22
Age, Customized [Count of Participants; unit: Participants]
  Age Category: 18-30 years | 0
  Age Category: 31-40 years | 2
  Age Category: 41-50 years | 1
  Age Category: 51-60 years | 6
  Age Category: 61-65 years | 1
  Age Category: 66-70 years | 0
  Age Category: Missing | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Waist Circumference [Mean (Full Range); unit: cm] — Population: On January 9, 2013, the field for waist circumference was removed as a required field in the database collection forms. As of that date, only 2 participants had records for waist circumference entered into the database.
  cm
    number analyzed (Participants) | 2
    (all) | 98.0 [95 to 101]
Weight [Mean (Full Range); unit: kg] — Population: On January 9, 2013, the field for weight was removed as a required field in the database collection forms. As of that date, only 6 participants had records for weight entered into the database.
  kg
    number analyzed (Participants) | 6
    (all) | 68.95 [57.1 to 78.1]
Height [Mean (Full Range); unit: cm] — Population: On January 9, 2013, the field for height was removed as a required field in the database collection forms. As of that date, only 6 participants had had records for height entered into the database.
  cm
    number analyzed (Participants) | 6
    (all) | 158.68 [132.0 to 170.5]
Parotid Fill Volume [Median (Full Range); unit: mL/min] — Fill volumes were determined by injecting saline using a syringe into the parotid. Injection was terminated when the parotid volume was full or a maximum of 1 mL was injected. Population: Two participants in the Safety population were never randomized. These two participants were thus entered in the table as "not randomized"
  mL/min
    Parotid randomized to dexamethasone irrigation: number analyzed (Participants) | 9
    Parotid randomized to dexamethasone irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation | 1.0 [0.6 to 1.0]
    Parotid randomized to placebo irrigation: number analyzed (Participants) | 9
    Parotid randomized to placebo irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to placebo irrigation | 1.0 [0.7 to 1.0]
    Not randomized, right-side parotid: number analyzed (Participants) | 2
    Not randomized, right-side parotid: number analyzed (parotid glands) | 2
    Not randomized, right-side parotid | 0.875 [0.75 to 1.00]
    Not randomized, left-side parotid: number analyzed (Participants) | 2
    Not randomized, left-side parotid: number analyzed (parotid glands) | 2
    Not randomized, left-side parotid | 0.875 [0.75 to 1.00]
Saliva Flow [Mean (Standard Deviation); unit: mL/min] — Population: Two participants in the safety population were not randomized and thus their saliva flow was not recorded at their baseline randomization visit.
  mL/min
    number analyzed (Participants) | 9
    number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation | 0.21250 (0.158850)
    Parotid randomized to placebo irrigation | 0.19096 (0.136399)
Focus Score [Median (Full Range); unit: score on a scale] — Focus score is the number of mononuclear cell infiltrates containing at least 50 inflammatory cells in a 4 mm² glandular section. Focus scores ≥1 are key criteria used in the diagnosis of inflammation in the oral component of Sjögren's Syndrome. Higher numbers are associated with more inflammation. (Range 0-12). Population: The biopsy to determine the Focus score was only performed on the right-side parotid, thus only half the parotids have focus scores at baseline (4 dexamethasone randomized parotids; 4 placebo randomized parotids). Three parotids (participants) did not have biopsies at baseline (Stage I Screening).
  score on a scale
    number analyzed (Participants) | 4
    number analyzed (parotid glands) | 4
    Parotid randomized to dexamethasone irrigation | 2.5 [1 to 12]
    Parotid randomized to placebo irrigation | 1.5 [0 to 2]
MRI Scan Evaluation [Count of Units; unit: parotid glands] — Baseline table counts are the count of parotid glands (2 per participant). In the table: "Abnormal, not clinically significant" is abbreviated as "Abnormal ncs"; "Abnormal, clinically significant" is abbreviated as "Abnormal cs". Population: Two participants in the Safety population were never randomized. The left and right parotids for these 2 participants were thus entered in the table as "not randomized"
  parotid glands
    Parotid randomized to dexamethasone irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation: Normal | 5
    Parotid randomized to dexamethasone irrigation: Abnormal ncs | 4
    Parotid randomized to dexamethasone irrigation: Abnormal cs | 0
    Parotid randomized to dexamethasone irrigation: Not done | 0
    Parotid randomized to placebo irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to placebo irrigation: Normal | 5
    Parotid randomized to placebo irrigation: Abnormal ncs | 4
    Parotid randomized to placebo irrigation: Abnormal cs | 0
    Parotid randomized to placebo irrigation: Not done | 0
    Not randomized, right-side parotid: number analyzed (parotid glands) | 2
    Not randomized, right-side parotid: Normal | 0
    Not randomized, right-side parotid: Abnormal ncs | 0
    Not randomized, right-side parotid: Abnormal cs | 0
    Not randomized, right-side parotid: Not done | 2
    Not randomized, left-side parotid: number analyzed (parotid glands) | 2
    Not randomized, left-side parotid: Normal | 0
    Not randomized, left-side parotid: Abnormal ncs | 0
    Not randomized, left-side parotid: Abnormal cs | 0
    Not randomized, left-side parotid: Not done | 2
Technetium Scan Evaluation [Count of Units; unit: parotid glands] — Baseline table counts are the count of parotid glands (2 per participant) Population: Two participants in the Safety population were never randomized. The left and right parotids for these 2 participants were thus entered in the table as "not randomized"
  parotid glands
    Parotid randomized to dexamethasone irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation: Normal | 4
    Parotid randomized to dexamethasone irrigation: Abnormal | 5
    Parotid randomized to dexamethasone irrigation: Not done | 0
    Placebo randomized parotid: Normal: number analyzed (parotid glands) | 9
    Placebo randomized parotid: Normal: Normal | 4
    Placebo randomized parotid: Normal: Abnormal | 5
    Placebo randomized parotid: Normal: Not done | 0
    Not randomized, right-side parotid: number analyzed (parotid glands) | 2
    Not randomized, right-side parotid: Normal | 0
    Not randomized, right-side parotid: Abnormal | 1
    Not randomized, right-side parotid: Not done | 1
    Not randomized, left-side parotid: number analyzed (parotid glands) | 2
    Not randomized, left-side parotid: Normal | 0
    Not randomized, left-side parotid: Abnormal | 1
    Not randomized, left-side parotid: Not done | 1
Technetium Isotope Uptake [Count of Units; unit: parotid glands] — Baseline table counts are the count of parotid glands (2 per participant). Population: Two participants in the Safety population were never randomized. The left and right parotids for these 2 participants were thus entered in the table as "not randomized"
  parotid glands
    Parotid randomized to dexamethasone irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation: Yes | 9
    Parotid randomized to dexamethasone irrigation: No | 0
    Parotid randomized to dexamethasone irrigation: Not done | 0
    Parotid randomized to placebo irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to placebo irrigation: Yes | 9
    Parotid randomized to placebo irrigation: No | 0
    Parotid randomized to placebo irrigation: Not done | 0
    Not randomized, right-side parotid: number analyzed (parotid glands) | 2
    Not randomized, right-side parotid: Yes | 1
    Not randomized, right-side parotid: No | 0
    Not randomized, right-side parotid: Not done | 1
    Not randomized, left-side parotid: number analyzed (parotid glands) | 2
    Not randomized, left-side parotid: Yes | 1
    Not randomized, left-side parotid: No | 0
    Not randomized, left-side parotid: Not done | 1
Technetium Release with Stimulation [Count of Units; unit: parotid glands] — Baseline table counts are the count of parotid glands (2 per participant). Population: Two participants in the Safety population were never randomized. The left and right parotids for these 2 participants were thus entered in the table as "not randomized"
  parotid glands
    Parotid randomized to dexamethasone irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to dexamethasone irrigation: Yes | 8
    Parotid randomized to dexamethasone irrigation: No | 1
    Parotid randomized to dexamethasone irrigation: Not done | 0
    Parotid randomized to placebo irrigation: number analyzed (parotid glands) | 9
    Parotid randomized to placebo irrigation: Yes | 7
    Parotid randomized to placebo irrigation: No | 2
    Parotid randomized to placebo irrigation: Not done | 0
    Not randomized, right-side parotid: number analyzed (parotid glands) | 2
    Not randomized, right-side parotid: Yes | 1
    Not randomized, right-side parotid: No | 0
    Not randomized, right-side parotid: Not done | 1
    Not randomized, left-side parotid: number analyzed (parotid glands) | 2
    Not randomized, left-side parotid: Yes | 1
    Not randomized, left-side parotid: No | 0
    Not randomized, left-side parotid: Not done | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Parotid Salivary Flow From Baseline (Day 0) to Day 56.
Description: Saliva flow rate was determined by weighing the saliva flow collected separately from each parotid (dexamethasone irrigated and placebo irrigated parotid) within a participant and dividing by collection time. Saliva was collected using a Teflon collection cup placed over the parotid duct orifice and held in place by slight negative pressure. Collection time was 1 minute. The primary outcome measure is looking at change from baseline at Study Day 56 and not the flow at any particular time.
Time Frame: Baseline (Study Day 0) to Study Day 56
Population: Primary Efficacy Population (PEP): all enrolled participants who receive all parotid irrigations on study Days 0 and 28, have the same treatment applied to the same parotid (regardless of random assignment) at both visits, and have values for the primary endpoint (i.e., change in salivary flow from Day 0 to Day 56).
Measure: Mean (Standard Error); unit: g/min
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
g/min | -0.01120 (0.049063) | -0.05204 (0.032029)
Statistical Analysis 1: Comparison: Dexamethasone Irrigation of Parotid Gland vs Placebo Irrigation of Parotid Gland; The mixed models analysis included all time points but it failed to converge. Therefore, an alternative analysis was performed using a paired t-test. Because the Satterthwaite correction [that was specified in the statistical analysis plan (SAP) for the mixed model] is not available for the paired t-test, it was not performed on the paired t-test. The final analysis was based upon the raw non-transformed saliva flow rates, as these measures were appropriate for the model used; Test type: Superiority — The standard deviation (SD) of the change in salivary flow was assumed to be 0.0168 for the placebo and 0.0906 for the dexamethasone parotid. The within-subject correlation between two glands was assumed to be 0.15. A total of 16 patients would be required to have 80% power to detect a one-sided 40% increase in dexamethasone-irrigated parotid glands compared with the saline irrigated parotid glands with respect to change in salivary flow from Day 0 to Day 56; p = 0.236, one-sided Paired t-test — No corrections were made for multiple comparisons because there was only one primary hypothesis

2. Secondary Outcome: Change in Parotid Salivary Flow From Baseline (Study Day 0) to Study Day 14.
Description: Saliva flow rate was determined by weighing the saliva flow collected separately from each parotid (dexamethasone irrigated and placebo irrigated parotid) within a participant and dividing by collection time. Saliva was collected using a Teflon collection cup placed over the parotid duct orifice and hel in place by slight negative pressure. Collection time was 1 minute. The outcome measure is looking at change from baseline at Study Day 14 and not the flow at any particular time.
Time Frame: Baseline to 14 days post-baseline
Population: Secondary Efficacy Population (SEP): all enrolled participants who receive at least one on-treatment set of parotid irrigations and have at least one salivary flow assessment after study Day 0.
Measure: Mean (Standard Error); unit: g/min
Units Other Than Participants: Parotid gland from one side of the mouth
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Number analyzed (Parotid gland from one side of the mouth) | 9 | 9
g/min | -0.01106 (0.075004) | 0.01875 (0.047825)
Statistical Analysis 1: Comparison: Dexamethasone Irrigation of Parotid Gland vs Placebo Irrigation of Parotid Gland; The mixed models analysis (including all time points: study days 14, 28, 42, 56) failed to converge; thus, an alternative analysis, as stated in the Statistical Analysis Plan, was performed using the paired t-test. The Satterthwaite correction (Statistical Analysis Plan) is not available for the paired t-test and was not performed on the paired t-test. The final analysis was based upon the raw non-transformed saliva flow rates since this statistical model achieved the best fit to the data; Test type: Superiority; p = 0.662, one-sided paired t-test

3. Secondary Outcome: Change in Parotid Salivary Flow From Baseline (Day 0) to Day 28.
Description: Saliva flow rate was determined by weighing the saliva flow collected separately from each parotid (dexamethasone irrigated and placebo irrigated parotid) within a participant and dividing by collection time. Saliva was collected using a Teflon collection cup placed over the parotid duct orifice and hel in place by slight negative pressure. Collection time was 1 minute. The outcome measure is looking at change from baseline at Study Day 28 and not the flow at any particular time.
Time Frame: Baseline to 28 days post-baseline
Population: as for outcome 2
Measure: Mean (Standard Error); unit: g/min
Units Other Than Participants: Parotid gland on one side of the mouth
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Number analyzed (Parotid gland on one side of the mouth) | 9 | 9
g/min | -0.09808 (0.058960) | -0.06678 (0.071649)
Statistical Analysis 1: Comparison: Dexamethasone Irrigation of Parotid Gland vs Placebo Irrigation of Parotid Gland; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.607, one-sided paired t-test

4. Secondary Outcome: Change in Parotid Salivary Flow From Baseline (Day 0) to Day 42.
Description: Saliva flow rate was determined by weighing the saliva flow collected separately from each parotid (dexamethasone irrigated and placebo irrigated parotid) within a participant and dividing by collection time. Saliva was collected using a Teflon collection cup placed over the parotid duct orifice and hel in place by slight negative pressure. Collection time was 1 minute. The outcome measure is looking at change from baseline at Study Day 42 and not the flow at any particular time.
Time Frame: Baseline to 42 days post-baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/min
Units Other Than Participants: Parotid galnd on one side of the mouth
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Number analyzed (Parotid galnd on one side of the mouth) | 9 | 9
g/min | 0.00224 (0.055472) | 0.01192 (0.031049)
Statistical Analysis 1: Comparison: Dexamethasone Irrigation of Parotid Gland vs Placebo Irrigation of Parotid Gland; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.586, one-sided paired t-test

5. Secondary Outcome: Patient Dry Mouth Questionnaire. Question: Do You Have More Difficulty Chewing Your Food Since Starting the Study?
Description: The questionnaire's question is on the whole participant level rather than on the individual parotid level; thus, no treatment group comparisons are possible. Possible responses: Yes or No.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Dexamethasone and Placebo Parotid Irrigation Groups are not applicable; Not measured by Body Side.
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 3
  Stage II Screening: No | 6
  Study Day 14: Yes | 1
  Study Day 14: No | 8
  Study Day 28: Yes | 2
  Study Day 28: No | 7
  Study Day 42: Yes | 1
  Study Day 42: No | 8
  Study Day 56: Yes | 2
  Study Day 56: No | 7

6. Secondary Outcome: Patient Dry Mouth Questionnaire. Question: If You Have More Difficulty Chewing Your Food Since Starting the Study, Why?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: number analyzed (Participants) | 3
  Stage II Screening: Pain | 0
  Stage II Screening: Dryness | 3
  Stage II Screening: Weakness | 0
  Stage II Screening: Too few Teeth | 0
  Stage II Screening: Other | 0
  Study Day 14: number analyzed (Participants) | 1
  Study Day 14: Pain | 0
  Study Day 14: Dryness | 1
  Study Day 14: Weakness | 0
  Study Day 14: Too few Teeth | 0
  Study Day 14: Other | 0
  Study Day 28: number analyzed (Participants) | 2
  Study Day 28: Pain | 0
  Study Day 28: Dryness | 2
  Study Day 28: Weakness | 0
  Study Day 28: Too few Teeth | 0
  Study Day 28: Other | 0
  Study Day 42: number analyzed (Participants) | 1
  Study Day 42: Pain | 0
  Study Day 42: Dryness | 1
  Study Day 42: Weakness | 0
  Study Day 42: Too few Teeth | 0
  Study Day 42: Other | 0
  Study Day 56: number analyzed (Participants) | 2
  Study Day 56: Pain | 0
  Study Day 56: Dryness | 2
  Study Day 56: Weakness | 0
  Study Day 56: Too few Teeth | 0
  Study Day 56: Other | 0

7. Secondary Outcome: Patient Dry Mouth Questionnaire. Question: Have You Experienced Any Changes in Your Sense of Smell Since Starting the Study?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 0
  Stage II Screening: No | 9
  Study Day 14: Yes | 0
  Study Day 14: No | 9
  Study Day 28: Yes | 0
  Study Day 28: No | 9
  Study Day 42: Yes | 0
  Study Day 42: No | 9
  Study Day 56: Yes | 0
  Study Day 56: No | 9

8. Secondary Outcome: Patient Dry Mouth Questionnaire: Have You Experienced Any Changes in Your Sense of Taste Since Starting the Study?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 1
  Stage II Screening: No | 8
  Study Day 14: Yes | 2
  Study Day 14: No | 7
  Study Day 28: Yes | 1
  Study Day 28: No | 8
  Study Day 42: Yes | 0
  Study Day 42: No | 9
  Study Day 56: Yes | 0
  Study Day 56: No | 9

9. Secondary Outcome: Patient Dry Mouth Questionnaire: If You Have Experienced Any Changes in Your Sense of Taste Since Starting the Study, Specify:
Description: The questionnaire's question is on the whole participant level rather than on the individual parotid level; thus, no treatment group comparisons are possible.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: number analyzed (Participants) | 1
  Stage II Screening: Foods taste different than they used to | 0
  Stage II Screening: Foods taste less intense (for example, less sweet) | 0
  Stage II Screening: Foods taste more intense (for example, more sweet) | 1
  Stage II Screening: I have persistent bad taste in my mouth | 0
  Study Day 14: number analyzed (Participants) | 2
  Study Day 14: Foods taste different than they used to | 0
  Study Day 14: Foods taste less intense (for example, less sweet) | 1
  Study Day 14: Foods taste more intense (for example, more sweet) | 1
  Study Day 14: I have persistent bad taste in my mouth | 0
  Study Day 28: number analyzed (Participants) | 1
  Study Day 28: Foods taste different than they used to | 1
  Study Day 28: Foods taste less intense (for example, less sweet) | 0
  Study Day 28: Foods taste more intense (for example, more sweet) | 0
  Study Day 28: I have persistent bad taste in my mouth | 0
  Study Day 42: number analyzed (Participants) | 0
  Study Day 42: Foods taste different than they used to | 0
  Study Day 42: Foods taste less intense (for example, less sweet) | 0
  Study Day 42: Foods taste more intense (for example, more sweet) | 0
  Study Day 42: I have persistent bad taste in my mouth | 0
  Study Day 56: number analyzed (Participants) | 0
  Study Day 56: Foods taste different than they used to | 0
  Study Day 56: Foods taste less intense (for example, less sweet) | 0
  Study Day 56: Foods taste more intense (for example, more sweet) | 0
  Study Day 56: I have persistent bad taste in my mouth | 0

10. Secondary Outcome: Patient Dry Mouth Questionnaire: Do You Have Any More Pain or Burning in Your Mouth or Head and Neck Region Since Starting the Study?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Dexamethasone and Placebo Parotid Irrigation Groups are not applicable; Not measured by Body Side.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 2
  Stage II Screening: No | 7
  Study Day 14: Yes | 2
  Study Day 14: No | 7
  Study Day 28: Yes | 1
  Study Day 28: No | 8
  Study Day 42: Yes | 1
  Study Day 42: No | 8
  Study Day 56: Yes | 1
  Study Day 56: No | 8

11. Secondary Outcome: Patient Dry Mouth Questionnaire: If You Have Any More Pain or Burning in Your Mouth or Head and Neck Region Since Starting the Study, Specify:
Description: as for outcome 9
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: number analyzed (Participants) | 2
  Stage II Screening: Mouth or tongue burns | 1
  Stage II Screening: I have tooth pain | 0
  Stage II Screening: I have gum pain | 0
  Stage II Screening: I have pain in my jaws or TMJ | 1
  Study Day 14: number analyzed (Participants) | 2
  Study Day 14: Mouth or tongue burns | 1
  Study Day 14: I have tooth pain | 0
  Study Day 14: I have gum pain | 0
  Study Day 14: I have pain in my jaws or TMJ | 1
  Study Day 28: number analyzed (Participants) | 1
  Study Day 28: Mouth or tongue burns | 0
  Study Day 28: I have tooth pain | 0
  Study Day 28: I have gum pain | 0
  Study Day 28: I have pain in my jaws or TMJ | 1
  Study Day 42: number analyzed (Participants) | 1
  Study Day 42: Mouth or tongue burns | 1
  Study Day 42: I have tooth pain | 0
  Study Day 42: I have gum pain | 0
  Study Day 42: I have pain in my jaws or TMJ | 0
  Study Day 56: number analyzed (Participants) | 1
  Study Day 56: Mouth or tongue burns | 0
  Study Day 56: I have tooth pain | 0
  Study Day 56: I have gum pain | 0
  Study Day 56: I have pain in my jaws or TMJ | 1

12. Secondary Outcome: Patient Dry Mouth Questionnaire: Do You Use Anything to Keep Your Mouth Moist?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 8
  Stage II Screening: No | 1
  Study Day 14: Yes | 9
  Study Day 14: No | 0
  Study Day 28: Yes | 9
  Study Day 28: No | 0
  Study Day 42: Yes | 9
  Study Day 42: No | 0
  Study Day 56: Yes | 8
  Study Day 56: No | 1

13. Secondary Outcome: Patient Dry Mouth Questionnaire: If You Use Something to Keep Your Mouth Moist, Specify:
Description: as for outcome 9
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline: Sip water | 8
  Baseline: Sip liquids other than water | 6
  Baseline: use commercial products | 4
  Baseline: Chew sugared gum or mints | 1
  Baseline: Chew sugarless gum or mints | 2
  Study Day 14: Sip water | 8
  Study Day 14: Sip liquids other than water | 6
  Study Day 14: use commercial products | 3
  Study Day 14: Chew sugared gum or mints | 1
  Study Day 14: Chew sugarless gum or mints | 4
  Study Day 28: Sip water | 8
  Study Day 28: Sip liquids other than water | 7
  Study Day 28: use commercial products | 4
  Study Day 28: Chew sugared gum or mints | 2
  Study Day 28: Chew sugarless gum or mints | 3
  Study Day 42: Sip water | 7
  Study Day 42: Sip liquids other than water | 5
  Study Day 42: use commercial products | 3
  Study Day 42: Chew sugared gum or mints | 2
  Study Day 42: Chew sugarless gum or mints | 3
  Study Day 56: Sip water | 8
  Study Day 56: Sip liquids other than water | 3
  Study Day 56: use commercial products | 3
  Study Day 56: Chew sugared gum or mints | 1
  Study Day 56: Chew sugarless gum or mints | 2

14. Secondary Outcome: Patient Dry Mouth Questionnaire: Does Your Mouth Feel More Dry When You Eat a Meal Since Starting the Study?
Description: The questionnaire's question is on the whole participant level rather than on the individual parotid level; thus, no treatment group comparisons are possible. Possible responses: Yes; No; Not sure.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 1
  Stage II Screening: No | 6
  Stage II Screening: Not Sure | 2
  Study Day 14: Yes | 1
  Study Day 14: No | 7
  Study Day 14: Not Sure | 1
  Study Day 28: Yes | 2
  Study Day 28: No | 7
  Study Day 28: Not Sure | 0
  Study Day 42: Yes | 1
  Study Day 42: No | 8
  Study Day 42: Not Sure | 0
  Study Day 56: Yes | 1
  Study Day 56: No | 7
  Study Day 56: Not Sure | 1

15. Secondary Outcome: Patient Dry Mouth Questionnaire: Does Your Mouth Feel More Dry Other Times of the Day Since Starting the Study?
Description: as for outcome 14
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 3
  Stage II Screening: No | 6
  Stage II Screening: Not Sure | 0
  Study Day 14: Yes | 5
  Study Day 14: No | 3
  Study Day 14: Not Sure | 1
  Study Day 28: Yes | 3
  Study Day 28: No | 5
  Study Day 28: Not Sure | 1
  Study Day 42: Yes | 2
  Study Day 42: No | 5
  Study Day 42: Not Sure | 2
  Study Day 56: Yes | 2
  Study Day 56: No | 6
  Study Day 56: Not Sure | 1

16. Secondary Outcome: Patient Dry Mouth Questionnaire: Does the Amount of Saliva in Your Mouth Most of the Time Seem to be:
Description: The questionnaire's question is on the whole participant level rather than on the individual parotid level; thus, no treatment group comparisons are possible. Possible responses: To little; to much; Do not notice it.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Too little | 4
  Stage II Screening: Too much | 0
  Stage II Screening: Do not notice it | 5
  Study Day 14: Too little | 6
  Study Day 14: Too much | 0
  Study Day 14: Do not notice it | 3
  Study Day 28: Too little | 5
  Study Day 28: Too much | 0
  Study Day 28: Do not notice it | 4
  Study Day 42: Too little | 5
  Study Day 42: Too much | 0
  Study Day 42: Do not notice it | 4
  Study Day 56: Too little | 4
  Study Day 56: Too much | 0
  Study Day 56: Do not notice it | 5

17. Secondary Outcome: Patient Dry Mouth Questionnaire: Do You Have More Difficulty Swallowing Dry Foods Without Additional Liquids Since Starting the Study?
Description: as for outcome 5
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Stage II Screening: Yes | 1
  Stage II Screening: No | 8
  Study Day 14: Yes | 1
  Study Day 14: No | 8
  Study Day 28: Yes | 3
  Study Day 28: No | 6
  Study Day 42: Yes | 3
  Study Day 42: No | 6
  Study Day 56: Yes | 1
  Study Day 56: No | 8

18. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: More Difficulty Chewing Food?
Description: Shift table with respect to the change from the Stage II Screening Visit (used as Baseline) for Study Days: 14, 28, 42, and 56
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 1
  Study Day 14: Screening II: Yes; Study Day: No | 2
  Study Day 14: Screening II: No; Study Day: Yes | 0
  Study Day 14: Screening II: No; Study Day: No | 6
  Study Day 28: Screening II: Yes; Study Day: Yes | 1
  Study Day 28: Screening II: Yes; Study Day: No | 2
  Study Day 28: Screening II: No; Study Day: Yes | 1
  Study Day 28: Screening II: No; Study Day: No | 5
  Study Day 42: Screening II: Yes; Study Day: Yes | 1
  Study Day 42: Screening II: Yes; Study Day: No | 2
  Study Day 42: Screening II: No; Study Day: Yes | 0
  Study Day 42: Screening II: No; Study Day: No | 6
  Study Day 56: Screening II: Yes; Study Day: Yes | 2
  Study Day 56: Screening II: Yes; Study Day: No | 1
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 6
Statistical Analysis 1: Comparison: Overall Study; McNemar's test on the study Day 14 shift table. The null hypothesis assumes the probability of subjects shifting from "yes" at Screening to "no" at Study Day 14 are equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 14. Alternative hypothesis is that probability of subjects shifting from "yes" at Screening to "no" at Study Day 14 is not equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 14; Test type: Other; p = 0.500, McNemar
Statistical Analysis 2: Comparison: Overall Study; McNemar's test on the study Day 28 shift table. The null hypothesis assumes the probability of subjects shifting from "yes" at Screening to "no" at Study Day 28 is equal to the probability of subjects shifting their answer from "no" at Screening to "yes" at Study Day 28. Alternative hypothesis is that probability of subjects shifting from "yes" at Screening to "no" at Study Day 28 is not equal to the probability of subjects shifting their answer from "no" at Screening to "yes" at Study Day 28; Test type: Other; p = 1.000, McNemar
Statistical Analysis 3: Comparison: Overall Study; McNemar's test on the study Day 42 shift table. The null hypothesis assumes the probability of subjects shifting from "yes" at Screening to "no" at Study Day 42 are equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 42. Alternative hypothesis is that probability of subjects shifting from "yes" at Screening to "no" at Study Day 42 is not equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 42; Test type: Other; p = 0.500, McNemar
Statistical Analysis 4: Comparison: Overall Study; McNemar's test on the study Day 56 shift table. The null hypothesis assumes the probability of subjects shifting from "yes" at Screening to "no" at Study Day 56 are equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 56. Alternative hypothesis is that probability of subjects shifting from "yes" at Screening to "no" at Study Day 56 is not equal to the probability of subjects shifting from "no" at Screening to "yes" at Study Day 56; Test type: Other; p = 1.000, McNemar

19. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Changes in Sense of Smell?
Description: Shift table with respect to the change from the Stage II Screening Visit (used as Baseline) for Study Days: 14, 28, 42, and 56. The shift table data were not sufficiently distributed to permit analysis with McNemar's test on any of the study days.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 0
  Study Day 14: Screening II: Yes; Study Day: No | 0
  Study Day 14: Screening II: No; Study Day: Yes | 0
  Study Day 14: Screening II: No; Study Day: No | 9
  Study Day 28: Screening II: Yes; Study Day: Yes | 0
  Study Day 28: Screening II: Yes; Study Day: No | 0
  Study Day 28: Screening II: No; Study Day: Yes | 0
  Study Day 28: Screening II: No; Study Day: No | 9
  Study Day 42: Screening II: Yes; Study Day: Yes | 0
  Study Day 42: Screening II: Yes; Study Day: No | 0
  Study Day 42: Screening II: No; Study Day: Yes | 0
  Study Day 42: Screening II: No; Study Day: No | 9
  Study Day 56: Screening II: Yes; Study Day: Yes | 0
  Study Day 56: Screening II: Yes; Study Day: No | 0
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 9

20. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Changes in Sense of Taste?
Description: Shift table with respect to the change from the Stage II Screening Visit (used as Baseline) for Study Days: 14, 28, 42, and 56. The shift table data were not sufficiently distributed to permit analysis with McNemar's test on Study Days 42 and 56.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 1
  Study Day 14: Screening II: Yes; Study Day: No | 0
  Study Day 14: Screening II: No; Study Day: Yes | 1
  Study Day 14: Screening II: No; Study Day: No | 7
  Study Day 28: Screening II: Yes; Study Day: Yes | 0
  Study Day 28: Screening II: Yes; Study Day: No | 1
  Study Day 28: Screening II: No; Study Day: Yes | 1
  Study Day 28: Screening II: No; Study Day: No | 7
  Study Day 42: Screening II: Yes; Study Day: Yes | 0
  Study Day 42: Screening II: Yes; Study Day: No | 1
  Study Day 42: Screening II: No; Study Day: Yes | 0
  Study Day 42: Screening II: No; Study Day: No | 8
  Study Day 56: Screening II: Yes; Study Day: Yes | 0
  Study Day 56: Screening II: Yes; Study Day: No | 1
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 8
Statistical Analysis 1: Comparison: Overall Study; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 2: Comparison: Overall Study; [analysis description as in outcome 18, analysis 2]; Test type: Other; p = 1.000, McNemar

21. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Pain/Burning in Mouth or Head/Neck?
Description: as for outcome 18
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 1
  Study Day 14: Screening II: Yes; Study Day: No | 1
  Study Day 14: Screening II: No; Study Day: Yes | 1
  Study Day 14: Screening II: No; Study Day: No | 6
  Study Day 28: Screening II: Yes; Study Day: Yes | 1
  Study Day 28: Screening II: Yes; Study Day: No | 1
  Study Day 28: Screening II: No; Study Day: Yes | 0
  Study Day 28: Screening II: No; Study Day: No | 7
  Study Day 42: Screening II: Yes; Study Day: Yes | 1
  Study Day 42: Screening II: Yes; Study Day: No | 1
  Study Day 42: Screening II: No; Study Day: Yes | 0
  Study Day 42: Screening II: No; Study Day: No | 7
  Study Day 56: Screening II: Yes; Study Day: Yes | 1
  Study Day 56: Screening II: Yes; Study Day: No | 1
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 7
Statistical Analysis 1: Comparison: Overall Study; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 2: Comparison: Overall Study; [analysis description as in outcome 18, analysis 2]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 3: Comparison: Overall Study; [analysis description as in outcome 18, analysis 3]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 4: Comparison: Overall Study; [analysis description as in outcome 18, analysis 4]; Test type: Other; p = 1.000, McNemar

22. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Use Anything to Keep Mouth Moist?
Description: as for outcome 19
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 8
  Study Day 14: Screening II: Yes; Study Day: No | 0
  Study Day 14: Screening II: No; Study Day: Yes | 1
  Study Day 14: Screening II: No; Study Day: No | 0
  Study Day 28: Screening II: Yes; Study Day: Yes | 8
  Study Day 28: Screening II: Yes; Study Day: No | 0
  Study Day 28: Screening II: No; Study Day: Yes | 1
  Study Day 28: Screening II: No; Study Day: No | 0
  Study Day 42: Screening II: Yes; Study Day: Yes | 8
  Study Day 42: Screening II: Yes; Study Day: No | 0
  Study Day 42: Screening II: No; Study Day: Yes | 1
  Study Day 42: Screening II: No; Study Day: No | 0
  Study Day 56: Screening II: Yes; Study Day: Yes | 8
  Study Day 56: Screening II: Yes; Study Day: No | 0
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 1

23. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Mouth Feel More Dry When You Eat?
Description: as for outcome 19
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: Secondary Efficacy Population (SEP): all enrolled participants who receive at least one on-treatment set of parotid irrigations and have at least one salivary flow assessment after study Day 0. The shift tables were limited to binary outcomes; participants that answered "not sure" were excluded from the shift tables.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: number analyzed (Participants) | 6
  Study Day 14: Screening II: Yes; Study Day: Yes | 1
  Study Day 14: Screening II: Yes; Study Day: No | 0
  Study Day 14: Screening II: No; Study Day: Yes | 0
  Study Day 14: Screening II: No; Study Day: No | 5
  Study Day 28: number analyzed (Participants) | 7
  Study Day 28: Screening II: Yes; Study Day: Yes | 1
  Study Day 28: Screening II: Yes; Study Day: No | 0
  Study Day 28: Screening II: No; Study Day: Yes | 0
  Study Day 28: Screening II: No; Study Day: No | 6
  Study Day 42: number analyzed (Participants) | 7
  Study Day 42: Screening II: Yes; Study Day: Yes | 1
  Study Day 42: Screening II: Yes; Study Day: No | 0
  Study Day 42: Screening II: No; Study Day: Yes | 0
  Study Day 42: Screening II: No; Study Day: No | 6
  Study Day 56: number analyzed (Participants) | 6
  Study Day 56: Screening II: Yes; Study Day: Yes | 1
  Study Day 56: Screening II: Yes; Study Day: No | 0
  Study Day 56: Screening II: No; Study Day: Yes | 0
  Study Day 56: Screening II: No; Study Day: No | 5

24. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Mouth Feel More Dry Other Times of Day?
Description: as for outcome 18
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: number analyzed (Participants) | 8
  Study Day 14: Screening II: Yes; Study Day: Yes | 2
  Study Day 14: Screening II: Yes; Study Day: No | 0
  Study Day 14: Screening II: No; Study Day: Yes | 3
  Study Day 14: Screening II: No; Study Day: No | 3
  Study Day 28: number analyzed (Participants) | 8
  Study Day 28: Screening II: Yes; Study Day: Yes | 1
  Study Day 28: Screening II: Yes; Study Day: No | 1
  Study Day 28: Screening II: No; Study Day: Yes | 2
  Study Day 28: Screening II: No; Study Day: No | 4
  Study Day 42: number analyzed (Participants) | 7
  Study Day 42: Screening II: Yes; Study Day: Yes | 1
  Study Day 42: Screening II: Yes; Study Day: No | 0
  Study Day 42: Screening II: No; Study Day: Yes | 1
  Study Day 42: Screening II: No; Study Day: No | 5
  Study Day 56: number analyzed (Participants) | 8
  Study Day 56: Screening II: Yes; Study Day: Yes | 1
  Study Day 56: Screening II: Yes; Study Day: No | 1
  Study Day 56: Screening II: No; Study Day: Yes | 1
  Study Day 56: Screening II: No; Study Day: No | 5
Statistical Analysis 1: Comparison: Overall Study; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 0.250, McNemar
Statistical Analysis 2: Comparison: Overall Study; [analysis description as in outcome 18, analysis 2]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 3: Comparison: Overall Study; [analysis description as in outcome 18, analysis 3]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 4: Comparison: Overall Study; [analysis description as in outcome 18, analysis 4]; Test type: Other; p = 1.000, McNemar

25. Secondary Outcome: Patient Dry Mouth Questionnaire Shift Table. Question: Difficulty Swallowing Dry Foods Without Liquids?
Description: as for outcome 18
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Screening II: Yes; Study Day: Yes | 0
  Study Day 14: Screening II: Yes; Study Day: No | 1
  Study Day 14: Screening II: No; Study Day: Yes | 1
  Study Day 14: Screening II: No; Study Day: No | 7
  Study Day 28: Screening II: Yes; Study Day: Yes | 0
  Study Day 28: Screening II: Yes; Study Day: No | 1
  Study Day 28: Screening II: No; Study Day: Yes | 3
  Study Day 28: Screening II: No; Study Day: No | 5
  Study Day 42: Screening II: Yes; Study Day: Yes | 1
  Study Day 42: Screening II: Yes; Study Day: No | 0
  Study Day 42: Screening II: No; Study Day: Yes | 2
  Study Day 42: Screening II: No; Study Day: No | 6
  Study Day 56: Screening II: Yes; Study Day: Yes | 0
  Study Day 56: Screening II: Yes; Study Day: No | 1
  Study Day 56: Screening II: No; Study Day: Yes | 1
  Study Day 56: Screening II: No; Study Day: No | 7
Statistical Analysis 1: Comparison: Overall Study; [analysis description as in outcome 18, analysis 1]; Test type: Other; p = 1.000, McNemar
Statistical Analysis 2: Comparison: Overall Study; [analysis description as in outcome 18, analysis 2]; Test type: Other; p = 0.625, McNemar
Statistical Analysis 3: Comparison: Overall Study; [analysis description as in outcome 18, analysis 3]; Test type: Other; p = 0.5000, McNemar
Statistical Analysis 4: Comparison: Overall Study; [analysis description as in outcome 18, analysis 4]; Test type: Other; p = 1.000, McNemar

26. Secondary Outcome: Sjögren's Disease Activity Index: Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient (Ordinal Numeric Scale)
Description: Ordinal Scale 0:least to 10:greatest level of disease activity
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 9
units on a scale
  Baseline | 5 [4 to 7]
  Study Day 14 | 5 [4 to 7]
  Study Day 28 | 5 [4 to 7]
  Study Day 42 | 5 [5 to 7]
  Study Day 56 | 5 [5 to 7]

27. Secondary Outcome: Sjögren's Disease Activity Index: Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient (Nominal Scale)
Description: Nominal scale values: Inactive; Low; Moderate; High
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline: Inactive | 0
  Baseline: Low | 2
  Baseline: Moderate | 7
  Baseline: High | 0
  Study Day 14: Inactive | 0
  Study Day 14: Low | 2
  Study Day 14: Moderate | 7
  Study Day 14: High | 0
  Study Day 28: Inactive | 0
  Study Day 28: Low | 2
  Study Day 28: Moderate | 7
  Study Day 28: High | 0
  Study Day 42: Inactive | 0
  Study Day 42: Low | 3
  Study Day 42: Moderate | 6
  Study Day 42: High | 0
  Study Day 56: Inactive | 0
  Study Day 56: Low | 4
  Study Day 56: Moderate | 5
  Study Day 56: High | 0

28. Secondary Outcome: Sjögren's Disease Activity Index: Do You Consider Your Patient in a Satisfactory State of 'Minimal Disease Activity'?
Description: Response: Yes or No
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline: Yes | 0
  Baseline: No | 9
  Study Day 14: Yes | 0
  Study Day 14: No | 9
  Study Day 28: Yes | 0
  Study Day 28: No | 9
  Study Day 42: Yes | 0
  Study Day 42: No | 9
  Study Day 56: Yes | 0
  Study Day 56: No | 9

29. Secondary Outcome: Sjögren's Disease Activity Index: Indicate the Level of Disease Activity in This Patient, Taking Into Account the Symptoms of Your Patient's (Dryness, Pain, Physical and Mental Fatigue), Ordinal Scores
Description: Ordinal Scale 0: least to 10: greatest level of disease activity.
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 9
score on a scale
  Baseline | 5 [5 to 7]
  Study Day 14 | 5 [5 to 7]
  Study Day 28 | 5 [5 to 7]
  Study Day 42 | 5 [5 to 7]
  Study Day 56 | 5 [4 to 7]

30. Secondary Outcome: Sjögren's Disease Activity Index: Compared With Baseline, This Participant's Primary Sjögren's Syndrome (pSS) Activity is Now:
Description: Nominal Scale: Much better; Better; The same; Worse; Much worse
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline: Much better | 0
  Baseline: Better | 0
  Baseline: The same | 7
  Baseline: Worse | 2
  Baseline: Much worse | 0
  Study Day 14: Much better | 0
  Study Day 14: Better | 0
  Study Day 14: The same | 7
  Study Day 14: Worse | 2
  Study Day 14: Much worse | 0
  Study Day 28: Much better | 0
  Study Day 28: Better | 0
  Study Day 28: The same | 7
  Study Day 28: Worse | 2
  Study Day 28: Much worse | 0
  Study Day 42: Much better | 0
  Study Day 42: Better | 0
  Study Day 42: The same | 9
  Study Day 42: Worse | 0
  Study Day 42: Much worse | 0
  Study Day 56: Much better | 0
  Study Day 56: Better | 1
  Study Day 56: The same | 8
  Study Day 56: Worse | 0
  Study Day 56: Much worse | 0

31. Secondary Outcome: Sjögren's Disease Activity Index: Compared With Baseline, do You Consider Your Patient Presents a Systemic Flare of the Participant's pSS (Primary Sjögren's Syndrome):
Description: Response: Yes; No
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline: Yes | 1
  Baseline: No | 8
  Study 14: Yes | 2
  Study 14: No | 7
  Study Day 28: Yes | 2
  Study Day 28: No | 7
  Study Day 42: Yes | 0
  Study Day 42: No | 9
  Study Day 56: Yes | 0
  Study Day 56: No | 9

32. Secondary Outcome: Sjögren's Disease Activity Index Shift Table. Question: Do You Consider Your Patient in a Satisfactory State of "Minimal Disease Activity? The Shift Table Data Was Not Rich Enough to Perform McNemar's Test on the Shift Tables of Any of the Study Days.
Description: Possible Response: Yes or No
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Yes | 0
  Study Day 14: No | 9
  Study Day 28: Yes | 0
  Study Day 28: No | 9
  Study Day 42: Yes | 0
  Study Day 42: No | 9
  Study Day 56: Yes | 0
  Study Day 56: No | 9

33. Secondary Outcome: Sjörgen's Disease Activity Index, Shift Table of Disease Activity Based on Patient's Symptoms From Baseline to Study Day 14 , Ordinal Scores
Description: Ordinal Scale 0: least to 10: greatest level of disease activity. Only cells in the shift table with participant counts greater than 0 are listed.
Time Frame: Baseline (Study Day 0) through Study Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=5; Study Day 14 SDAI=5 | 4
  Baseline SDAI=5; Study Day 14 SDAI=6 | 1
  Baseline SDAI=6; Study Day 14 SDAI=5 | 1
  Baseline SDAI=6; Study Day 14 SDAI=6 | 1
  Baseline SDAI=6; Study Day 14 SDAI=7 | 1
  Baseline SDAI=7; Study Day 14 SDAI=7 | 1

34. Secondary Outcome: Sjörgen's Disease Activity Index, Shift Table of Disease Activity Based on Patient's Symptoms From Baseline to Study Day 28 , Ordinal Scores
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) through Study Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=5; Study Day 28 SDAI=5 | 4
  Baseline SDAI=5; Study Day 28 SDAI=6 | 1
  Baseline SDAI=6; Study Day 28 SDAI=5 | 2
  Baseline SDAI=6; Study Day 28 SDAI=7 | 1
  Baseline SDAI=7; Study Day 28 SDAI=7 | 1

35. Secondary Outcome: Sjörgen's Disease Activity Index, Shift Table of Disease Activity Based on Patient's Symptoms From Baseline to Study Day 42 , Ordinal Scores
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) through Study Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=5; Study Day 42 SDAI=5 | 4
  Baseline SDAI=5; Study Day 42 SDAI=6 | 1
  Baseline SDAI=6; Study Day 42 SDAI=5 | 1
  Baseline SDAI=6; Study Day 42 SDAI=6 | 2
  Baseline SDAI=7; Study Day 42 SDAI=7 | 1

36. Secondary Outcome: Sjörgen's Disease Activity Index, Shift Table of Disease Activity Based on Patient's Symptoms From Baseline to Study Day 56 , Ordinal Scores
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=5; Study Day 56 SDAI=4 | 1
  Baseline SDAI=5; Study Day 56 SDAI=5 | 3
  Baseline SDAI=5; Study Day 56 SDAI=6 | 1
  Baseline SDAI=6; Study Day 56 SDAI=5 | 2
  Baseline SDAI=6; Study Day 56 SDAI=6 | 1
  Baseline SDAI=7; Study Day 56 SDAI=7 | 1

37. Secondary Outcome: Sjörgen's Disease Activity Index (SDAI): Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient (Nominal Scale) the Shift From Baseline to the Given Study Day, Nominal Scale
Description: Possible response on nominal scale: Inactive; Low; Moderate; High SDAI.
Time Frame: Baseline (Study Day 0) to Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Study Day 14: Baseline Inactive to Study Day Inactive | 0
  Study Day 14: Baseline Inactive to Study Day Low | 0
  Study Day 14: Baseline Inactive to Study Day Moderate | 0
  Study Day 14: Baseline Inactive to Study Day High | 0
  Study Day 14: Baseline Low to Study Day Inactive | 0
  Study Day 14: Baseline Low to Study Day Low | 2
  Study Day 14: Baseline Low to Study Day Moderate | 0
  Study Day 14: Baseline Low to Study Day High | 0
  Study Day 14: Baseline Moderate to Study Day Inactive | 0
  Study Day 14: Baseline Moderate to Study Day Low | 0
  Study Day 14: Baseline Moderate to Study Day Moderate | 7
  Study Day 14: Baseline Moderate to Study Day High | 0
  Study Day 14: Baseline High to Study Day Inactive | 0
  Study Day 14: Baseline High to Study Day Low | 0
  Study Day 14: Baseline High to Study Day Moderate | 0
  Study Day 14: Baseline High to Study Day High | 0
  Study Day 28: Baseline Inactive to Study Day Inactive | 0
  Study Day 28: Baseline Inactive to Study Day Low | 0
  Study Day 28: Baseline Inactive to Study Day Moderate | 0
  Study Day 28: Baseline Inactive to Study Day High | 0
  Study Day 28: Baseline Low to Study Day Inactive | 0
  Study Day 28: Baseline Low to Study Day Low | 2
  Study Day 28: Baseline Low to Study Day Moderate | 0
  Study Day 28: Baseline Low to Study Day High | 0
  Study Day 28: Baseline Moderate to Study Day Inactive | 0
  Study Day 28: Baseline Moderate to Study Day Low | 0
  Study Day 28: Baseline Moderate to Study Day Moderate | 7
  Study Day 28: Baseline Moderate to Study Day High | 0
  Study Day 28: Baseline High to Study Day Inactive | 0
  Study Day 28: Baseline High to Study Day Low | 0
  Study Day 28: Baseline High to Study Day Moderate | 0
  Study Day 28: Baseline High to Study Day High | 0
  Study Day 42: Baseline Inactive to Study Day Inactive | 0
  Study Day 42: Baseline Inactive to Study Day Low | 0
  Study Day 42: Baseline Inactive to Study Day Moderate | 0
  Study Day 42: Baseline Inactive to Study Day High | 0
  Study Day 42: Baseline Low to Study Day Inactive | 0
  Study Day 42: Baseline Low to Study Day Low | 2
  Study Day 42: Baseline Low to Study Day Moderate | 0
  Study Day 42: Baseline Low to Study Day High | 0
  Study Day 42: Baseline Moderate to Study Day Inactive | 0
  Study Day 42: Baseline Moderate to Study Day Low | 1
  Study Day 42: Baseline Moderate to Study Day Moderate | 6
  Study Day 42: Baseline Moderate to Study Day High | 0
  Study Day 42: Baseline High to Study Day Inactive | 0
  Study Day 42: Baseline High to Study Day Low | 0
  Study Day 42: Baseline High to Study Day Moderate | 0
  Study Day 42: Baseline High to Study Day High | 0
  Study Day 56: Baseline Inactive to Study Day Inactive | 0
  Study Day 56: Baseline Inactive to Study Day Low | 0
  Study Day 56: Baseline Inactive to Study Day Moderate | 0
  Study Day 56: Baseline Inactive to Study Day High | 0
  Study Day 56: Baseline Low to Study Day Inactive | 0
  Study Day 56: Baseline Low to Study Day Low | 2
  Study Day 56: Baseline Low to Study Day Moderate | 0
  Study Day 56: Baseline Low to Study Day High | 0
  Study Day 56: Baseline Moderate to Study Day Inactive | 0
  Study Day 56: Baseline Moderate to Study Day Low | 2
  Study Day 56: Baseline Moderate to Study Day Moderate | 5
  Study Day 56: Baseline Moderate to Study Day High | 0
  Study Day 56: Baseline High to Study Day Inactive | 0
  Study Day 56: Baseline High to Study Day Low | 0
  Study Day 56: Baseline High to Study Day Moderate | 0
  Study Day 56: Baseline High to Study Day High | 0

38. Secondary Outcome: Sjörgen's Disease Activity Index (SDAI): Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient the Shift From Baseline to Study Day 14, Ordinal Scale
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) to Study Day 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=4; Study Day 14 SDAI=4 | 1
  Baseline SDAI=5; Study Day 14 SDAI=5 | 4
  Baseline SDAI=6; Study Day 14 SDAI=5 | 2
  Baseline SDAI=6; Study Day 14 SDAI=7 | 1
  Baseline SDAI=7; Study Day 14 SDAI=7 | 1

39. Secondary Outcome: Sjörgen's Disease Activity Index (SDAI): Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient the Shift From Baseline to Study Day 28, Ordinal Scale
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) to Study Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=4; Study Day 28 SDAI=4 | 1
  Baseline SDAI=5; Study Day 28 SDAI=5 | 4
  Baseline SDAI=6; Study Day 28 SDAI=5 | 2
  Baseline SDAI=6; Study Day 28 SDAI=7 | 1
  Baseline SDAI=7; Study Day 28 SDAI=7 | 1

40. Secondary Outcome: Sjörgen's Disease Activity Index (SDAI): Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient the Shift From Baseline to Study Day 42, Ordinal Scale
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) to Study Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=4; Study Day 42 SDAI=5 | 1
  Baseline SDAI=5; Study Day 42 SDAI=5 | 4
  Baseline SDAI=6; Study Day 42 SDAI=5 | 3
  Baseline SDAI=7; Study Day 42 SDAI=7 | 1

41. Secondary Outcome: Sjörgen's Disease Activity Index (SDAI): Indicate, According to Your Clinical Experience, the Level of Disease Activity in This Patient the Shift From Baseline to Study Day 56, Ordinal Scale
Description: as for outcome 33
Time Frame: Baseline (Study Day 0) to Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 9
Participants
  Baseline SDAI=4; Study Day 56 SDAI=5 | 1
  Baseline SDAI=5; Study Day 56 SDAI=5 | 4
  Baseline SDAI=6; Study Day 56 SDAI=5 | 3
  Baseline SDAI=7; Study Day 56 SDAI=7 | 1

42. Secondary Outcome: Summary Statistics of MRI Scans
Description: Medical evaluations of MRI Scans. Possible evaluations include: i) Normal; ii) Abnormal, not clinically significant; iii) Abnormal, clinically significant.
Time Frame: Stage II Screening (within 6 wks before Baseline (Study Day 0)) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Participants
  Stage II Screening Visit: MRI Normal | 5 | 5
  Stage II Screening Visit: MRI Abnormal, not clinically signficant | 4 | 4
  Stage II Screening Visit: MRI Abnormal, clinically signficant | 0 | 0
  Study Day 56: MRI Normal | 5 | 6
  Study Day 56: MRI Abnormal, not clinically signficant | 3 | 3
  Study Day 56: MRI Abnormal, clinically signficant | 1 | 0

43. Secondary Outcome: Shift Table of the Change in Parotid MRI at Study Day 56 From Stage II Screening Visit
Description: Change in the evaluations of the parotid MRI scans at Study Day 56 from Stage II Screening Visit. Possible MRI evaluations at both Baseline and Study Day 56 include: i)Normal; ii) Abnormal, not clinically significant (Abnormal ncs); and iii) Abnormal, clinically significant (Abnormal cs).
Time Frame: Stage II Screening (within 6 wks before Baseline (Study Day 0)) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Participants
  Screening Normal; Study Day 56 Normal | 4 | 5
  Screening Normal; Study Day 56 Abnormal ncs | 0 | 0
  Screening Normal; Study Day 56 Abnormal cs | 1 | 0
  Screening Abnormal ncs; Study Day 56 Normal | 1 | 1
  Screening Abnormal ncs; Study Day 56 Abnormal ncs | 3 | 3
  Screening Abnormal ncs; Study Day 56 Abnormal cs | 0 | 0
  Screening Abnormal cs; Study Day 56 Normal | 0 | 0
  Screening Abnormal cs; Study Day 56 Abnormal ncs | 0 | 0
  Screening Abnormal cs; Study Day 56 Abnormal cs | 0 | 0

44. Secondary Outcome: Summary Statistics of Technetium Scans
Description: Medical evaluations of Technetium Scans. Possible evaluations include: i) Normal; and ii) Abnormal.
Time Frame: Stage II Screening (within 6 wks before Baseline (Study Day 0)) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Participants
  Stage II Screening Visit: Normal | 4 | 4
  Stage II Screening Visit: Abnormal | 5 | 5
  Study Day 56: Normal | 4 | 5
  Study Day 56: Abnormal | 5 | 4

45. Secondary Outcome: Shift Table of the Change in Parotid Technetium Scan at Study Day 56 From Stage II Screening Visit
Description: Change in the evaluations of the parotid technetium scans at Study Day 56 from Stage II Screening Visit. Possible technetium scan evaluations at both Baseline and Study Day 56 include: Normal; Abnormal.
Time Frame: Stage II Screening (within 6 wks before Baseline (Study Day 0)) through Study Day 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 9 | 9
Participants
  Screening Normal; Study Day 56 Normal | 4 | 4
  Baseline Normal; Study Day 56 Abnormal | 0 | 0
  Baseline Abnormal; Study Day 56 Normal | 0 | 1
  Baseline Abnormal; Study Day 56 Abnormal | 5 | 4

46. Secondary Outcome: Summary Statistics of Focus Score
Description: Focus score is the number of mononuclear cell infiltrates containing at least 50 inflammatory cells in a 4 mm² glandular section. Focus scores ≥1 are key criteria used in the diagnosis of inflammation in the oral component of Sjögren's Syndrome. Higher numbers are associated with more inflammation. (Range 0-12).
Time Frame: Stage II screening (within 6 wks before baseline) through 56 days post-baseline
Population: Secondary Efficacy Population (SEP). Since only the right parotid was biopsied, 9 parotids were biopsied (5 dexamethasone and 4 placebo randomized parotids). At Screening only 4/5 dexamethasone and 4/4 placebo randomized parotids were biopsied. At Study Day 56 only 3/5 dexamethasone and 4/4 placebo randomized parotids were biopsied.
Measure: Median (Full Range); unit: score on a scale
Units Other Than Participants: Parotid gland on right side of mouth
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 4 | 4
Number analyzed (Parotid gland on right side of mouth) | 4 | 4
score on a scale
  Stage II Screening | 2.5 [1 to 12] | 1.5 [0 to 2]
  Study Day 56: number analyzed (Participants) | 3 | 4
  Study Day 56: number analyzed (Parotid gland on right side of mouth) | 3 | 4
  Study Day 56 | 1 [0 to 3] | 0.5 [0 to 5]

47. Secondary Outcome: Shift Table of Focus Scores From Stage II Screening to Study Day 56
Description: Focus score is the number of mononuclear cell infiltrates containing at least 50 inflammatory cells in a 4 mm² glandular section. Table data are the shift in focus score from Stage II Screening to Study Day 56. Only shift table cells with more than 0 participants were included in the Outcome Measure Data Table below.
Time Frame: Stage II Screening (within 6 wks before baseline) through 56 days post-baseline
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Irrigation of Parotid Gland | Placebo Irrigation of Parotid Gland
Number analyzed (Participants) | 5 | 4
Participants
  Screening Focus=0; Day 56 Focus=0 | 0 | 1
  Screening Focus=1; Day 56 Focus=1 | 1 | 1
  Screening Focus=2; Day 56 Focus=0 | 1 | 1
  Screening Focus=2; Day 56 Focus=5 | 0 | 1
  Screening Focus=3; Day 56 Focus=not done | 1 | 0
  Screening Focus=12; Day 56 Focus=3 | 1 | 0
  Screening Focus=not done; Day 56 Focus=not done | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (AEs) are being reported in this document. Reporting period was 71 days from Randomization (Study Day 0) through Safety Follow-up (71 days).
Description: Adverse events were graded according to a descriptive scale based on the NIAID Division of Acquired Immunodeficiency Syndrome Table for Grading the Severity of Adverse Events. Adverse events were summarized by parotid treatment when related to the side of the mouth of parotid irrigation; otherwise, adverse events were summarized as not related to side of the mouth.
Groups:
- Dexamethasone Irrigation: Adverse event from the side of the mouth that received the parotid dexamethasone irrigation
- Placebo Irrigation: Adverse event from the side of the mouth that received the parotid placebo irrigation
- Side of Mouth Not Applicable: Side of mouth is not applicable to the adverse event
Arm/Group | Dexamethasone Irrigation | Placebo Irrigation | Side of Mouth Not Applicable
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/9 | 2/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Irrigation (N=9) | Placebo Irrigation (N=9) | Side of Mouth Not Applicable (N=9)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Elevated liver enzymes (ALT, AST)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Migraine Headache
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — Vertigo
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ecchymosis right side of face

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT01316770/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT01316770/SAP_001.pdf